CLINICAL TRIAL: NCT04564950
Title: Influence of Periodontitis and Coronary Heart Disease on Galectin-3 in Serum and Saliva
Brief Title: Influence of Periodontitis and Coronary Heart Disease on Galectin-3
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Principal Investigator, University of Messina
Other Study IDs: 18-16-2018
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Observation of salivary Galectin-3 levels and correlation of salivary Galectin -3 evels with periodontal disease
  Interventions: Other: Observation of serum and salivary Galectin-3 levels
- Periodontitis: Observation of salivary Galectin-3 levels and correlation of salivary Galectin -3 evels with periodontal disease
  Interventions: Other: Observation of serum and salivary Galectin-3 levels
- Coronary heart disease: Observation of salivary Galectin-3 levels and correlation of salivary Galectin -3 evels with periodontal disease
  Interventions: Other: Observation of serum and salivary Galectin-3 levels
- Coronary heart disease + periodontitis: Observation of salivary Galectin-3 levels and correlation of salivary Galectin -3 evels with periodontal disease
  Interventions: Other: Observation of serum and salivary Galectin-3 levels

INTERVENTIONS:
Other: Observation of serum and salivary Galectin-3 levels — Observation of serum and salivary Galectin-3 levels and correlation with periodontal indices

SUMMARY:
The aim of this study was to analyze the association between serum and salivary Galectin-3 levels in patients with periodontitis. Furthermore, the objective was to determine if the periodontitis influenced serum and salivary Galectin-3 levels

DETAILED DESCRIPTION:
Healthy controls (n=38), patients with CHD (n=39), periodontitis (n=40), and a combination of periodontitis + CHD (n=38) were enrolled in the present study. The analyzed sample undergo a demographical, clinical and periodontal evaluation and serological analyses including Endothelin-1 (ET-1) and for serum and salivary Galectin-3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 16 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy controls (n=38), patients with CHD (n=39), periodontitis (n=40), and a combination of periodontitis + CHD (n=38)
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Changes of Clinical Attachment Level (mm) | 1-year
  Measurment of changes in Clinical Attachment Level

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Official website